CLINICAL TRIAL: NCT01425528
Title: Pilot Study to Assess Impact of Kuvan® Supplementation as an Adjunct Treatment in Subjects With Dominantly-inherited GTPCH Deficiency on Mood, Behavioral and Motor Phenotypes
Brief Title: Study of Kuvan Treatment in Adults With GTPCH Deficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 48052
Record Dates: First submitted 2011-08-25; First posted 2011-08-30 (Estimated); Results first posted 2014-04-08 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2014-03

CONDITIONS: GTP Cyclohydrolase Deficiency
MeSH Terms: interventions — sapropterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kuvan Cohort 1 (Experimental): This cohort will be enrolled first. Analysis will be done to determine the optimum dosing of Kuvan to normalize BH4 levels in the Cerebral Spinal Fluid. This cohort will begin at a dose of 20mg/kg/day.
  Interventions: Drug: Sapropterin
- Kuvan Cohort 2 (Experimental): Participants in cohort 2 will be enrolled after the analysis of cohort 1 data has taken place. Dosing for cohort 2 will be based on results obtained in cohort 1, but will plan on starting at 30 mg/kg/day.
  Interventions: Drug: Sapropterin

INTERVENTIONS:
Drug: Sapropterin — Sapropterin will be taken daily for 12 or 24 weeks. Starting dose will be 20mg/kg/day and will increase at the 8 week visit to 30 mg/kg/day. Dosing may be further increased to as high as 40 mg/kg/day in attempt to normalize BH4 levels in CSF. Starting dose for Cohort 2 will be determined from data analysis in Cohort 1.
  Other Names: Kuvan

SUMMARY:
The purpose of this study is to identify the dose of Kuvan needed to normalize the levels of tetrahydrobiopterin (BH4) in patients with a Guanosine Triphosphate Cyclohydrolase (GTPCH) deficiency and to asses the potential impact of oral Kuvan on mood and function in individuals with GTPCH deficiency who may be experiencing symptoms of anxiety, depression, fatigue, trouble concentrating, or memory loss. This will be a phase one study. The investigators will monitor patients over a period of three to six months while on the medication. Medication levels will be monitored by measuring the BH4 levels in cerebral spinal fluid (CSF). Patients will undergo a baseline lumbar puncture and two follow-up lumbar punctures for this purpose. The investigators will also monitor emotional function and motor function.

ELIGIBILITY:
Inclusion Criteria:

* established diagnosis of GTPCH deficiency, supported by appropriate family history, CSF neurotransmitter studies, skin fibroblast enzyme assay and/or mutation analysis
* minimum age 18 years
* identified by self or others to have symptoms of anxiety, depression, fatigue, or other neurocognitive dysfunction (trouble concentrating, memory loss, etc)
* willingness to undergo at least 2 CSF evaluations for BH4 and neurotransmitter levels over an 8 to 12 week period

Exclusion Criteria:

* age < 18 years old
* unwillingness to undergo repeated CSF analysis
* lack of supporting diagnostic criteria
* concomitant medical problems or medications which would increase risk of Kuvan®
* concomitant psychiatric state, such as severe depression with suicidal ideation that requires immediate referral and alternative treatment intervention
* prior history of back surgery, abnormality or chronic pain that in the opinion of the investigator would increase risks associated with lumbar puncture
* significant obesity that might increase difficulty or risk in performing lumbar puncture
* if female, unwillingness to use birth control during the period of study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn J Swoboda, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from August 2011 through August 2013. Participants were patients who had been seen clinically for GTPCH deficiency and indicated previously that they would be interested in future research.
Pre-assignment Details: This is a pilot study and all participants are in the treatment group.
Groups:
- Cohort 1: This cohort will be enrolled first. Analysis will be done to determine the optimum dosing of Kuvan to normalize BH4 levels in the Cerebral Spinal Fluid.
- Cohort 2: Participants in cohort 2 will be enrolled after the analysis of cohort 1 data has taken place. Dosing for cohort 2 will be based on results obtained in cohort 1.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 6 | 6
Completed | 5 | 5
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: This cohort will be enrolled first. Analysis will be done to determine the optimum dosing of Kuvan to normalize BH4 levels in the Cerebral Spinal Fluid.
  Sapropterin: Sapropterin will be taken daily for 12 or 24 weeks. Starting dose will be 20mg/kg/day and will increase at the 8 week visit to 30 mg/kg/day. Dosing may be further increased to as high as 40 mg/kg/day in attempt to normalize BH4 levels in CSF. Starting dose for Cohort 2 will be determined from data analysis in Cohort 1.
- Cohort 2: Participants in cohort 2 will be enrolled after the analysis of cohort 1 data has taken place. Dosing for cohort 2 will be based on results obtained in cohort 1.
  Sapropterin: Sapropterin will be taken daily for 12 or 24 weeks. Starting dose will be 20mg/kg/day and will increase at the 8 week visit to 30 mg/kg/day. Dosing may be further increased to as high as 40 mg/kg/day in attempt to normalize BH4 levels in CSF. Starting dose for Cohort 2 will be determined from data analysis in Cohort 1.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Full Range); unit: years] | 42 [29 to 62] | 28 [18 to 37] | 35 [18 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in BH4 Levels in Cerebral Spinal Fluid
Description: Identify dosing range of oral Kuvan® necessary and sufficient to normalize CSF BH4 levels in adults with GTPCH Deficiency.
Time Frame: Baseline, 8 wks, 12 wks
Population: Data from 4 of 6 participants was analyzed for Kuvan Cohort 1 and for Kuvan Cohort 2 for this outcome measure. 2 participant withdrew, 1 participant's diagnosis was reclassified and we were unable to obtain baseline CSF on 1 participant.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 4 | 4
nmol/L
  Change in BH4 from Baseline at 8 weeks | 6 (1.4) | 10.7 (4.8)
  Change in BH4 from Baseline at 12 weeks | 5.3 (3.8) | 13.2 (3.9)

ADVERSE EVENTS:
Time Frame: Per protocol, adverse event data was collected from Baseline visit to 24 week Extension Visit
Description: Any untoward or unfavorable medical occurrence in a human subject, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the subject's participation in the research, whether or not considered related to the subject's participation in the research
Arm/Group | Cohort 1 | Cohort 2
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=6)
Uncontrollable Anger (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=6)
Post LP Headache (General disorders) | 2 (2) | 3 (4)
Viral Illness (General disorders) | 2 (2) | 3 (3)
GI illness (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 2 (3) | 1 (1)
root canal (General disorders) | 1 (1) | 0 (0)
Limb Trauma (General disorders) | 0 (0) | 1 (1) — Sprained Ankle
Pain (General disorders) | 1 (1) | 2 (2) — Increase in baseline pain
Depression (General disorders) | 0 (0) | 1 (1) — Worsening of baseline depression

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes